CLINICAL TRIAL: NCT06915636
Title: A Randomized Face-to-face Comparative Study of Low-energy 1064nm Laser With Large Spot Size and DPL in the Treatment of Rosacea
Brief Title: Comparative Study of Low-Energy 1064nm Laser and DPL in Rosacea Treatment
Acronym: DPL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025007
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DPL (Experimental): Half of the face was randomly treated with DPL, with an energy of 6-8 J/cm2, at an interval of 10 days, for a total of 8 treatments.
  Interventions: Other: DPL
- Large spot low-energy 1064nm laser (Experimental): One randomly assigned half of the face was treated with a large-spot, low-energy 1064nm laser at an energy of 0.8-1 J/cm², administered at 10-day intervals, for a total of 8 treatment sessions.
  Interventions: Other: DPL

INTERVENTIONS:
Other: DPL — Half of the face was randomly treated with DPL, with an energy of 6-8 J/cm2, at an interval of 10 days, for a total of 8 treatments.One randomly assigned half of the face was treated with a large-spot, low-energy 1064nm laser at an energy of 0.8-1 J/cm², administered at 10-day intervals, for a total of 8 treatment sessions.

SUMMARY:
Rosacea is a common skin disease characterized by transient flushing or persistent erythema and vasodilation symptoms on the face. In more severe cases, papules and pustules may appear in the central part of the face. Rosacea can be classified into four subtypes based on clinical manifestations: erythematotelangiectatic type, papulopustular type, rhinophyma type, and ocular rosacea type. Although the pathophysiology of rosacea is not fully understood, it has been found in previous studies that it is related to abnormal neurovascular and immune responses to various stimuli. Since rosacea is essentially chronic and recurrent, its treatment is difficult and usually requires lifelong management through lifestyle changes. The treatment methods vary depending on the severity and clinical subtype. Facial flushing and telangiectasia are common symptoms of rosacea, and they respond well to laser treatment with wavelengths that selectively absorb oxyhemoglobin, such as pulsed dye laser (PDL), intense pulsed light (IPL), and long-pulse Nd:YAG. Alexandrite laser is widely used for pigmented skin lesions and hair removal due to its absorption characteristics within the melanin spectrum. Recently, there has been increasing interest in using Alexandrite laser for treating vascular lesions, especially deeper ones, as it is relatively easily absorbed by deoxyhemoglobin and can penetrate deeper into the dermis than PDL. However, so far, there is little evidence regarding the effectiveness of Alexandrite laser in treating rosacea. In Kim et al.'s only available randomized clinical trial to date, the authors reported that the effect of dual-wavelength Alexandrite/Nd:YAG treatment for rosacea was comparable to that of PDL.

The unique photothermal effect of the large-spot low-energy mode of 1064nm Q-switched Nd:YAG laser can enhance endogenous porphyrin activity, inhibit Propionibacterium acnes activity, penetrate deeper into the dermis to reach sebaceous glands, regulate sebum secretion, and promote inflammation absorption. Rosacea mainly presents as dilated capillaries and/or red patches, and this laser's wavelength is located in the peak absorption region of hemoglobin, which selectively absorbs oxyhemoglobin. According to the selective photothermal effect of light, it destroys capillaries and inhibits their formation, thereby promoting inflammation regression and achieving the purpose of preventing and treating post-inflammatory erythema after acne. In addition, its photothermal effect can also stimulate collagen regeneration, stimulate the rearrangement of collagen fibers and elastic fibers, repair the barrier, and reduce the formation of acne-induced depressed scars.

DPL is a single narrow-band IPL device that combines the dual advantages of PDL and IPL. Its wavelength range is 500-600 nm, covering two absorption peaks of oxyhemoglobin including 542 nm and 577 nm, achieving higher energy concentration, higher vascular selectivity, and more precise treatment. This also makes it more precise and efficient in treating superficial vascular lesions.

In this study, researchers conducted a randomized face-to-face comparison trial of large-spot low-energy 1064nm laser and DPL to explore their clinical efficacy and safety for rosacea and attempted to compare whether there are differences in clinical treatment between the two for rosacea. Participants were involved in the study to assess the outcomes.

DETAILED DESCRIPTION:
Rosacea is a common, chronic inflammatory skin disorder primarily affecting the face, characterized by episodic or persistent redness, visible blood vessels (vasodilation), and, in more severe cases, the development of pimples or pustules. The condition often begins with frequent flushing, particularly in response to triggers such as heat, stress, or certain foods. Over time, it may lead to more persistent erythema, particularly in the central areas of the face, which can have a significant cosmetic impact on patients. In the most advanced stages of rosacea, the skin may develop thickened areas, particularly around the nose, a condition known as rhinophyma. Rosacea can be classified into four subtypes based on its clinical presentation: erythematotelangiectatic, which is marked by redness and visible blood vessels; papulopustular, which resembles acne with the formation of pimples and pustules; rhinophyma, which involves skin thickening, particularly around the nose; and ocular rosacea, which affects the eyes and can lead to dryness, irritation, and in severe cases, vision impairment.

While the exact cause of rosacea is not fully understood, it is widely believed to involve a combination of genetic factors, environmental triggers, and abnormalities in the immune and neurovascular systems. Many studies suggest that rosacea patients may have heightened sensitivity to various external and internal stimuli, such as UV light, spicy foods, and temperature extremes. Additionally, there is evidence indicating that rosacea may be associated with dysregulation of the blood vessels in the face, resulting in frequent flushing and persistent redness. Other potential contributing factors include the overgrowth of the skin bacterium *Demodex* and inflammatory responses to certain microbes.

Given that rosacea is a lifelong condition that typically follows a relapsing-remitting course, managing the disease can be challenging. While there is no cure, treatments are available to control symptoms and minimize flare-ups. These treatments range from topical medications to laser therapies and lifestyle modifications. Patients are often advised to avoid known triggers, such as hot drinks, spicy foods, and environmental factors that might cause excessive flushing. Medical management usually includes topical or oral antibiotics, such as metronidazole or tetracycline, which can help reduce inflammation and control the appearance of pimples. However, because rosacea tends to be chronic, its management often requires long-term treatment, which can include laser therapy.

Laser treatment is one of the most effective options for addressing the vascular component of rosacea, such as visible blood vessels and facial redness. Lasers that specifically target oxyhemoglobin in blood vessels, such as pulsed dye laser (PDL), intense pulsed light (IPL), and long-pulse Nd:YAG lasers, have been shown to be effective at reducing erythema and telangiectasia. Alexandrite laser, traditionally used for the treatment of pigmented lesions and hair removal, has also gained attention for its potential in treating deeper vascular lesions in rosacea. This is due to its ability to penetrate deeper into the dermis and its selective absorption by deoxygenated hemoglobin, making it an attractive option for treating larger or deeper vascular lesions that may not respond well to other laser treatments. However, research on the efficacy of Alexandrite lasers specifically for rosacea treatment is still limited. The most significant randomized clinical trial available, conducted by Kim et al., found that dual-wavelength Alexandrite/Nd:YAG laser treatment was comparable to pulsed dye laser in its effectiveness for managing rosacea.

Another promising treatment option for rosacea is the 1064nm Q-switched Nd:YAG laser, which operates using a large spot and low-energy mode. This laser offers a unique photothermal effect that is particularly effective for treating the vascular components of rosacea. The laser can enhance the activity of endogenous porphyrins, which helps to inhibit the activity of *Propionibacterium acnes*, a bacterium associated with rosacea and acne. The 1064nm wavelength of the Nd:YAG laser is especially effective for targeting the dilated blood vessels that are a hallmark of rosacea. By selectively absorbing oxyhemoglobin, the laser can destroy blood vessels and inhibit their formation, leading to a reduction in redness and inflammation. Additionally, the laser's photothermal effect stimulates collagen regeneration, which helps to repair the skin's barrier, promote the rearrangement of collagen fibers, and reduce the formation of acne-induced scars. This makes it a comprehensive treatment not only for the vascular symptoms of rosacea but also for addressing some of the long-term cosmetic issues, such as scarring.

In addition to these established laser therapies, the use of DPL (dual pulsed light), a narrow-band intense pulsed light device, has also shown promise in treating rosacea. DPL combines the advantages of both PDL and IPL by delivering a more concentrated energy output in the range of 500-600 nm. This wavelength range includes key absorption peaks for oxyhemoglobin, specifically 542 nm and 577 nm, allowing for higher vascular selectivity and greater energy precision. As a result, DPL is particularly effective at targeting superficial vascular lesions and is a useful option for patients with more delicate or sensitive skin types. Its ability to precisely target blood vessels makes it an efficient treatment for rosacea with a minimal risk of side effects.

In this study, the researchers designed a randomized, face-to-face comparison trial to investigate the clinical efficacy and safety of two different treatment modalities for rosacea: the large-spot low-energy 1064nm Nd:YAG laser and the DPL device. The trial aimed to compare the effectiveness of these treatments in reducing the symptoms of rosacea, such as facial redness, visible blood vessels, and inflammation, as well as their impact on overall skin texture and appearance. By comparing these two approaches directly, the researchers sought to determine if one treatment offered superior results in terms of patient outcomes, safety, and long-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Those with a history of photosensitivity;
* Those who have combined with severe immunological diseases;
* Those with a tendency to form scars;
* Pregnant or lactating women;
* Alcoholics;
* Those with other facial disorders;
* Those with mental illness or mental disorders who cannot cooperate with treatment;
* During pregnancy or lactation;
* Those with serious internal medical diseases;
* Those with poor compliance or non-cooperation in mental disorders.

Exclusion Criteria:

* Age range: 18 - 60 years old, gender not limited;
* Patients diagnosed with rosacea in bilateral facial lesion areas with basically symmetrical distribution based on dermoscopy and clinical manifestations;
* Patients with good cognitive function and normal mental state;
* Patients with good communication skills;
* Patients who voluntarily participate in this study and sign the informed consent form.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2024-12-07 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
IGA score | Baseline level, six weeks, twelve weeks
  The IGA score can be used to estimate the overall severity of the patient's condition. The score ranges from 0 to 4, with higher scores indicating more severe conditions.

SECONDARY OUTCOMES:
CEA score | Baseline level, six weeks, twelve weeks
  The CEA score can be used to estimate the overall severity of the patient's condition. The score ranges from 0 to 4, with higher scores indicating more severe conditions.
GFSS score | Baseline level, six weeks, twelve weeks
  The name of the scale is Global Flushing Severity Scale. The score ranges from 0 to 4, with higher scores indicating more severe conditions.
patient satisfaction evaluation | twelve weeks
  Patient satisfaction was evaluated as very satisfied, satisfied, relatively satisfied and dissatisfied.
erythema index | Baseline level, six weeks, twelve weeks
  Use non-invasive skin analyzer to measure the erythema index on the patient's facial skin at each follow-up visit.The larger the value, the more severe the erythema.
Dermatology Life Quality Index score | Baseline level, twelve weeks
  The name of the scale is Dermatology Life Quality Index. It was used to assess the changes in quality of life before and after treatment. The Dermatology Life Quality Index score ranges from 0 to 29, with higher scores indicating a greater impact of the disease on the patient's quality of life.
transepidermal water loss | Baseline level, six weeks, twelve weeks
  Use non-invasive skin analyzer to measure the transepidermal water loss on the patient's facial skin at each follow-up visit.The larger the value, the more severe the transdermal water loss.
melanin index | Baseline level, six weeks, twelve weeks
  Use non-invasive skin analyzer to measure the melanin index on the patient's facial skin at each follow-up visit.The larger the value, the higher the melanin level.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong University, Xian, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ruan J, Zheng Y, Cai S. Efficacy and safety comparison between pulsed dye laser and intense pulsed light configured with different wavelength bands in treating erythematotelangiectatic rosacea. Lasers Med Sci. 2024 Jun 1;39(1):146. doi: 10.1007/s10103-024-04098-9. PMID 38822948
- [Result] Varughese N, Keller L, Goldberg DJ. Split-face comparison between single-band and dual-band pulsed light technology for treatment of photodamage. J Cosmet Laser Ther. 2016 Aug;18(4):213-6. doi: 10.1080/14764172.2016.1177188. PMID 27183026
- [Result] Fu Y, Quan Y, Zhao W, Liu Z, Peng J, Pang X, Zhao B, Tan L, Zhou Q, Shao L, Wang H, Hou S. Low-Energy Delicate Pulsed Light Therapy for Sensitive Skin: A Retrospective Study. J Cosmet Dermatol. 2025 Jan;24(1):e16781. doi: 10.1111/jocd.16781. PMID 39780466